CLINICAL TRIAL: NCT01215812
Title: Analysis of Cases of Sexual Assault in Taiwan
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 098013-3
Record Dates: First submitted 2010-10-05; First posted 2010-10-07 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2011-09

CONDITIONS: Sexual Assault

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
The aim of this study was to analyze victims, assailants, assaults, evidentiary examinations and treatment characteristics of cases of sexual assault sought emergency care at Far Eastern Memorial Hospital、National Cheng Kung University Hospital、Taoyuan General Hospital, Department of Health, Executive Tuan, R.O.C.、National Taiwan University Hospital Yun-Lin Branch、Hospital and National Taiwan University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* all cases

Exclusion Criteria:

* nil

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: sexual assault
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2009-08; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, Taiwan